CLINICAL TRIAL: NCT03964688
Title: Randomized Controlled Trial on the Effect of Vitamin C Supplementation in Autologous Stem Cell Transplantations
Brief Title: Effect of Vitamin C in Autologous Stem Cell Transplantations
Acronym: VICAST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL68010.068.18; 2018-004135-77 (EudraCT Number)
Record Dates: First submitted 2019-05-09; First posted 2019-05-28 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Myeloma Multiple; Lymphoma
Keywords: vitamin C; ascorbate; ascorbic acid; autologous stem cell transplantation
MeSH Terms: conditions — Multiple Myeloma; Lymphoma | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: double blind placebo-controlled randomized trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin C (Experimental): vitamin C intravenous during hospitalization, followed with vitamin C oral
  Interventions: Drug: Vitamin C
- Placebo (Experimental): placebo intravenous during hospitalization, followed with placebo oral
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Vitamin C — vitamin C intravenous during hospitalization, after oral, total 6 weeks.
  Other Names: ascorbic acid
  Arms: Vitamin C
Drug: Placebos — placebo intravenous during hospitalization, after oral, total 6 weeks
  Other Names: placebo
  Arms: Placebo

SUMMARY:
In the study the investigators will randomize patients that receive an autologous stem cell transplantation for myeloma or lymphoma for treatment with vitamin C or placebo during 6 weeks. Primary endpoint will be immune recovery.

DETAILED DESCRIPTION:
Rationale: Recent studies showed that ascorbic acid (AA) stimulates proliferation and maturation of T lymphocytes and natural killer (NK) cells. Chemotherapy results in depletion of those cells and thereby an increased infection rate. A pilot study showed low levels of AA in the plasma of several patients after chemotherapy followed by autologous stem cell transplantation for hematological malignancies. AA supplementation could be beneficial to the recovery of the immune system in these patients.

Objective: The aim of this study is to examine the effect of vitamin C supplementation on immune recovery in patients with autologous stem cell transplantation. The aim of the run-in phase of the study is to examine the effect of intravenous vitamin C supplementation on plasma concentrations of vitamin C in patients with autologous stem cell transplantation at day 14 in order to be sure that in the intervention study accurate AA plasma levels will be present.

Study design: run-in phase, followed by randomized controlled trial Study population: All participants will be adults (minimally 18 years old) that are planed to receive an autologous stem cell transplantation for multiple myeloma or lymphoma and are recruited at the MUMC+. In total there will be 3 expected (run-in phase) + 44 (randomized controlled trial) participants.

Main study parameters/endpoints: Primary endpoints will be AA plasma level on day 14 (run-in phase) and the day of neutrophil recovery after stem cell transplantation (randomized-controlled phase). Secondary endpoints will be AA leukocyte levels, infection rate, duration of hospital stay, side effects of chemotherapy, overall survival, coagulation parameters, platelet reactivity, fibrinolysis and quality of life.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

AA supplementation could be beneficial for the immune recovery in the participants of this study. The risks associated with participation in this study are low. Vitamin C supplementation is safe and hardly has any documented side effects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* written informed consent
* diagnosis of malignant lymphoma or multiple myeloma
* require chemotherapy plus autologous stem cell transplantation as standard of care for the disease at that stage
* central venous catheter in place or planned

Exclusion Criteria:

* inability to understand the nature and extent of the trial and the procedures required
* history of kidney stones
* kidney failure requiring dialysis or eGFR <30 mL/min. (CDK-EPI formula)
* history of G6PD deficiency
* life expectancy < 1 month
* use of immunosuppressive medication other than chemotherapy and corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
immune recovery | day 14-28
  the day of repopulation (return of neutrophil to at least 0.5 × 109/l) after autologous stem cell transplantation.

SECONDARY OUTCOMES:
AA plasma levels | day 14
  AA plasma levels
AA leukocyte levels | day 14
  AA leukocyte levels
Incidence of infections/ neutropenic fever | day 1-28
  fever and infections during hospitalization
Days of hospitalization | dag 1-28
  number of days patients are admitted in our hospital
Days with fever (≥ 38.5° C) | day 1-28
  Amount of days admitted patients have a fever
Incidence of bloodstream infections | day1-28
  number of bloodstream infections of admitted patients
Quality of life according to the EORTC QLQ-C30 | Day 0, day 14, day 42
  quality of live questionaire
Overall survival (3 months) | 3 months
  overall survival at 3 months
Relapse rates (3 months) | 3 months
  relapse rate at 3 months
Use of systemic antimicrobial agents (incidence and duration) | dau 1-28
  use of antibiotics during hospitalization
platelet reactivity | day 10
  platelet reactivity tests
ROS production | day 10
  ROS production platelets
platelet mitochondrial dysfunction | day 10
  platelet mitochondrial function test
number and severity of bleeding episodes during admission | day 1-28
  number and severity of bleeding episodes during admission

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Bos, Principal Investigator — Maastricht University Medical Center
Locations (1):
- MUMC+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No